CLINICAL TRIAL: NCT01888874
Title: Randomized, Double-blind, Placebo-controlled, Multicenter, Phase IIb Dose Finding Study of GLPG0634 Administered for 24 Weeks in Combination With Methotrexate to Subjects With Moderately to Severely Active Rheumatoid Arthritis Who Have an Inadequate Response to Methotrexate Alone
Brief Title: Dose-finding Study of GLPG0634 as add-on to Methotrexate in Active Rheumatoid Arthritis Participants (DARWIN1)
Acronym: DARWIN1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLPG0634-CL-203 (DARWIN1); 2012-003635-31 (EudraCT Number)
Record Dates: First submitted 2013-06-26; First posted 2013-06-28 (Estimated); Results first posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Methotrexate inadequate responders
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — GLPG0634

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Placebo (Placebo Comparator): Participants received GLPG0634 matching placebo capsules, orally, twice daily (BID) during Weeks 1 to 12. Participants who were responders (having at least 20 percent [%] improvement on TJC68 and SJC66) remained on placebo while nonresponders were re-randomized to GLPG0634 100 milligram (mg) once daily (QD) or 50 mg BID during Weeks 13 to 24.
  Interventions: Drug: Placebo
- GLPG0634 50 mg QD (Experimental): Participants received GLPG0634 50 mg capsules, orally, QD during Weeks 1 to 12. Participants who were responders (having at least 20% improvement on TJC68 and SJC66) remained on 50 mg QD while nonresponders were re-randomized to 100 mg QD during Weeks 13 to 24.
  Interventions: Drug: GLPG0634
- GLPG0634 100 mg QD (Experimental): Participants received GLPG0634 100 mg capsules, orally, QD during Weeks 1 to 24.
  Interventions: Drug: GLPG0634
- GLPG0634 200 mg QD (Experimental): Participants received GLPG0634 200 mg capsules, orally, QD during Weeks 1 to 24.
  Interventions: Drug: GLPG0634
- GLPG0634 25 mg BID (Experimental): Participants received GLPG0634 25 mg capsules, orally, BID during Weeks 1 to 12. Participants who were responders (having at least 20% improvement on TJC68 and SJC66) remained on 25 mg BID while nonresponders were re-randomized to 50 mg BID during Weeks 13 to 24.
  Interventions: Drug: GLPG0634
- GLPG0634 50 mg BID (Experimental): Participants received GLPG0634 50 mg capsules, orally, BID during Weeks 1 to 24.
  Interventions: Drug: GLPG0634
- GLPG0634 100 mg BID (Experimental): Participants received GLPG0634 100 mg capsules, orally, BID during Weeks 1 to 24.
  Interventions: Drug: GLPG0634

INTERVENTIONS:
Drug: GLPG0634 — GLPG0634 capsules.
  Arms: GLPG0634 100 mg BID; GLPG0634 100 mg QD; GLPG0634 200 mg QD; GLPG0634 25 mg BID; GLPG0634 50 mg BID; GLPG0634 50 mg QD
Drug: Placebo — Placebo capsules.
  Arms: Placebo

SUMMARY:
Participants suffering from active rheumatoid arthritis despite continued treatment with methotrexate were evaluated for improvement of disease activity (efficacy) when taking GLPG0634 (3 different doses - 50 milligram [mg], 100 mg and 200 mg daily -, each evaluated as once daily [QD] and twice daily [BID] regimen) or matching placebo for 24 weeks.

•During the course of the study, patients were also examined for any side effects that could occur (safety and tolerability), and the amount of GLPG0634 present in the blood (Pharmacokinetics) as well as the effects of GLPG0634 on disease- and mechanism of action-related parameters in the blood (Pharmacodynamics) were determined. Also, the effects of different doses and dose regiments of GLPG0634 administration on participants' disability, fatigue, and quality of life were evaluated.

DETAILED DESCRIPTION:
* Treatment duration was 24 weeks in total.
* However, at Week 12, participants on placebo who did not achieve a 20% improvement in swollen joint count(SJC66) and tender joint count (TJC68) were re-randomized (automatically via interactive voice/web response [IXRS]) to treatment to receive GLPG0634 100 mg QD or 50 mg BID doses in a blinded fashion, participants on 50 mg QD who had not achieved a 20% improvement in SJC66 and TJC68 were assigned to 100 mg QD and participants on 25 mg BID. who did not achieve a 20% improvement in SJC66 and TJC68 were assigned to 50 mg BID. All continued the study until Week 24.
* Participants in the other groups maintained their randomized treatment until Week 24.

ELIGIBILITY:
Inclusion Criteria:

* have a diagnosis of RA since at least 6 months and meeting the 2010 ACR/EULAR criteria of RA and ACR functional class I-III,
* have ≥6 swollen joints (from a 66 joint count) and ≥8 tender joints (from a 68 joint count) at Screening and at Baseline,
* Screening serum c-reactive protein ≥0.7 x upper limit of laboratory normal range (ULN),
* have received MTX for ≥6 months and have been on a stable dose (15 to 25 mg/week) of MTX for at least 4 weeks prior to Screening and willing to continue on their current regimen for the duration of the study. Stable doses of MTX as low as 10 mg/week are allowed when there is documented evidence of intolerance or safety issues at higher doses.

Exclusion Criteria:

* current therapy with any disease-modifying anti-rheumatic drugs (DMARD) other than MTX,
* current or previous RA treatment with a biologic DMARD, with the exception of biologic DMARDs administered in a single clinical study setting more than 6 months prior to Screening (12 months for rituximab or other B cell depleting agents), where the biologic DMARD was effective, and if discontinued, this should not be due to lack of efficacy,
* previous treatment at any time with a cytotoxic agent, other than MTX, before Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 599 (Actual)
Dates: Start 2013-07-17 (Actual); Primary Completion 2015-02-18 (Actual); Study Completion 2015-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Galapagos Study Director, Study Director — Galapagos NV
Locations (142):
- United States (28):
  - Rheumatology Associates of North Alabama, PC, Huntsville, Alabama
  - Artho Care, Arthritis Care & Research P.C., Gilbert, Arizona
  - Arizona Arthritis & Rheumatology Research PLLC, Phoenix, Arizona
  - C.V. Mehta MD Medical Corporation, Hemet, California
  - Center for Innovative TherapyDivision of Rheumatology, UCSD, La Jolla, California
  - Desert Medical Advances, Palm Desert, California
  - Desert Valley Medical Center, Victorville, California
  - Infosphere Clinical Research, Inc., West Hills, California
  - RASF Clinical Research Center, Boca Raton, Florida
  - Millennium Research, Ormond Beach, Florida
  - Lovelace Scientific Resources, Venice, Florida
  - Arthritis Center of North GA, Gainesville, Georgia
  - Idaho Arthritis Center, Meridian, Idaho
  - The Arthritis Center, Springfield, Illinois
  - Professional Research Network of Kansas, Wichita, Kansas
  - Arthritis Treatment Center, Frederick, Maryland
  - Klein and Associates MD, Hagerstown, Maryland
  - Private practice, Lansing, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Physicians East, Greenville, North Carolina
  - Health Research of Oklahoma, Oklahoma City, Oklahoma
  - Altoona Center Clinical Research, Duncansville, Pennsylvania
  - Austin Rheumatology Research PA, Austin, Texas
  - Arthritis Centers of Texas, Dallas, Texas
  - Pioneer Research Solutions Inc, Houston, Texas
  - Crossroads Clinical Research, LLC, Victoria, Texas
  - Seattle Rheumatology Associates, PLLC, Seattle, Washington
  - Mountain State Clinical Research, Clarksburg, West Virginia
- Argentina (6):
  - Atencion Integral en Reumatologa, Buenos Aires
  - Rheumatology OMI, Buenos Aires
  - Instituto Reumatologico, Córdoba
  - Instituto Medico CER, Quilmes
  - Instituto de Asistencia Reumatologia Integral, San Fernando
  - Centro Médico Privado de Reumatología, San Miguel de Tucumán
- Australia (4):
  - Royal Prince Alfred Hospital, Camperdown
  - Monash Medical Centre, Clayton
  - Repatriation General Hospital, Daw Park
  - Princess Alexandra Hospital, Woolloongabba
- Medical University/ AKH Vienna/ Dep.of Rheumatology 6J, Vienna, Austria
- Belgium (6):
  - Cliniques Universitaires St-Luc, Brussels
  - Hospital Brugmann, Brussels
  - Rheuma Instituut, Hasselt
  - AZ Groeninge, Kortrijk
  - UZ Leuven, Leuven
  - CHU de Liège, Liège
- Bulgaria (6):
  - "Multiprofile Hospital for Active Treatment - Kaspela" LTD, Plovdiv
  - MHAT Ruse AD, Rousse
  - Clinic of Rheumatology MHAT, Sofia
  - Diagnostic Consultative Center "Sveta Anna" LTD, Sofia
  - National Transport Hospital "Tsar Boris" III, Sofia
  - Rheumatology Clinic, Sofia
- Chile (6):
  - Hospital Regional "Guillermo Grant Benavente", Concepción
  - Instituto Terapias Oncologicas Providencia, Santiago
  - Prosalud, Santiago
  - Someal SA, Santiago
  - Centro de Investigacion Clínica del Sur Freire, Temuco
  - Private Office, Temuco
- Colombia (9):
  - Centro Integral de Reumatologia de Caribe, Barranquilla
  - Fundación del caribe para la investigación medica Fundación BIOS, Barranquilla
  - Centro Integral de Reumatologia e Inmunologia SAS, Bogotá
  - Cirei Sas, Bogotá
  - Idearg S.A.S., Bogotá
  - Medicity S.A.S., Bucaramanga
  - Clinica de Arthritis Temprana S.A.S., Cali
  - Preventive Care SAS, Cundinamarca
  - Hospital Pablo Tobon Uribe, Medellín
- Czechia (5):
  - Revmatologie S.R.O, Brno
  - Ambulance Revmatologie a Interniho Lekarstvi, Kladno
  - Revmatologicka ambulance, Praha-Nusle
  - Medical Plus, s.r.o., Uherské Hradiště
  - PV-Medical, Zlín
- Hopitaux universitaires de Strasbourg, Strasbourg, France
- Germany (5):
  - Charite Mitte, Rheumatologie Neue Therapien, Berlin
  - Schlossparkklinik - Akad. Lehrkrankenhaus Charite, Berlin
  - Klinikum Goethe-Universität, Frankfurt
  - Schwerpunktpraxis fuer Rheumatologie, Hamburg
  - Rheumazentrum Ruhrgebiet, Herne
- Guatemala (6):
  - Centro Medico, Guatemala City
  - Clinica de Especialidades Medicas, Guatemala City
  - Clinica Medica Especializada en Reumatologia, Guatemala City
  - Clinica Medica, Guatemala City
  - Reuma S.A., Guatemala City
  - Reuma-Centro, Guatemala City
- Hungary (7):
  - DRC, Balatonfüred
  - Budai Irgalmasrendi Korhaz, Budapest
  - Qualiclinic Ltd, Budapest
  - Revita Clinic, Budapest
  - Markhot Ferenc Korhaz, Eger
  - Bekes Megyei Pandy Kalman Korhaz, Reumatologiai Osztaly, Gyula
  - Csolnoky Ferenc County Hospital, Veszprém
- Israel (3):
  - Carmel Medical Center, Haifa
  - Rambam Medical Center, Haifa
  - Sheba Medical Center, Ramat Gan
- Latvia (5):
  - M&M Centre Ltd., Ādaži
  - Meda D, Daugavplis
  - L. Atikes doktorats, Liepāja
  - "Bruninieku" polyclinic, Riga
  - Arija's Ancane's Family Doctor, Riga
- Mexico (7):
  - Centro de Estudios de Investigacion Basica y Clinica, SC, Guadalajara
  - Arké Estudios Clínicos, México
  - Clinstile, S.A. de C.V., México
  - Hospital General de México, México
  - Accelerium Clinical Research, Monterrey
  - Hospital Universitario José E. González, Monterrey
  - Centro de Alta Especialidad en Reumatología e Investigación del Potosí, S.C., San Luis Potosí City
- IMSP Institutul de Cardiologie, Chisinau, Moldova
- New Zealand (3):
  - North Shore hospital, Auckland
  - Waikato Hospital, Hamilton
  - Timaru Rheumatology Studies, Timaru
- Poland (12):
  - NZOZ Osteo-Medic s.c., Bialystok
  - Silesiana Centrum Medyczne, Bytom
  - Medica Pro Familia Sp. z o.o. S.K.A., Katowice
  - Centrum Medyczne Plejady, Krakow
  - Nowomed, Krakow
  - Nzoz "Dobry Lekarz", Krakow
  - NZOZ Przychodnia Lekarska "Eskulap", Skierniewice
  - Powiatowy Zakrad Opieki Zdrowotnej w Starachowicach, Starachowice
  - NS ZOZ Medicus Bonus, Środa Wielkopolska
  - NZOZ Nasz Lekarz, Torun
  - AMED Medical Center, Warsaw
  - Wojewodzki Szpital Specjalistyczny we Wroclawiu, Wroclaw
- Russia (7):
  - I.M. Sechenov First Moscow State Medical University, Moscow
  - Research Institute of Rheumatology RAMS, Moscow
  - State University of Medicine and Dentistry, Moscow
  - City Clinical Hospital 5, Nizhny Novgorod
  - Ryazan State Medical University, Ryazan
  - City Hospital # 26, Saint Petersburg
  - Vladimir Reg Clin Hosp, Vladimir
- Spain (6):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Reina Sofa, Córdoba
  - Hospital General Universitario de Elche, Elche
  - Hospital Universitario de Mostoles, Móstoles
  - Consorci Sanitari Parc Tauli, Sabadell
  - Hospital Infanta Luisa, Seville
- Ukraine (8):
  - City Hospital #5, Donetsk
  - V. Gusak Institute of Urgent and Recovery Surgery, Donetsk
  - City Hospital #13, Kharkiv
  - City Hospital #8, Kharkiv
  - Government Institution, Kharkiv
  - Central Outpatient Hospital of Deanyanskyy Distric, Kiev
  - Central regional polyclinic of Pechersk District, Kyiv
  - Municipal Institution Lutsk City Clinical Hospital, Lutsk

REFERENCES:
- [Derived] Balsa A, Wassenberg S, Tanaka Y, Tournadre A, Orzechowski HD, Rajendran V, Lendl U, Stiers PJ, Watson C, Caporali R, Galloway J, Verschueren P. Effect of Filgotinib on Body Mass Index (BMI) and Effect of Baseline BMI on the Efficacy and Safety of Filgotinib in Rheumatoid Arthritis. Rheumatol Ther. 2023 Dec;10(6):1555-1574. doi: 10.1007/s40744-023-00599-1. Epub 2023 Sep 25. PMID 37747626
- [Derived] Combe B, Besuyen R, Gomez-Centeno A, Matsubara T, Sancho Jimenez JJ, Yin Z, Buch MH. Geographic Analysis of the Safety and Efficacy of Filgotinib in Rheumatoid Arthritis. Rheumatol Ther. 2023 Feb;10(1):35-51. doi: 10.1007/s40744-022-00494-1. Epub 2022 Oct 7. PMID 36205910
- [Derived] Tarrant JM, Galien R, Li W, Goyal L, Pan Y, Hawtin R, Zhang W, Van der Aa A, Taylor PC. Filgotinib, a JAK1 Inhibitor, Modulates Disease-Related Biomarkers in Rheumatoid Arthritis: Results from Two Randomized, Controlled Phase 2b Trials. Rheumatol Ther. 2020 Mar;7(1):173-190. doi: 10.1007/s40744-019-00192-5. Epub 2020 Jan 7. PMID 31912462
- [Derived] Westhovens R, Taylor PC, Alten R, Pavlova D, Enriquez-Sosa F, Mazur M, Greenwald M, Van der Aa A, Vanhoutte F, Tasset C, Harrison P. Filgotinib (GLPG0634/GS-6034), an oral JAK1 selective inhibitor, is effective in combination with methotrexate (MTX) in patients with active rheumatoid arthritis and insufficient response to MTX: results from a randomised, dose-finding study (DARWIN 1). Ann Rheum Dis. 2017 Jun;76(6):998-1008. doi: 10.1136/annrheumdis-2016-210104. Epub 2016 Dec 19. PMID 27993829

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Europe, South America, North America, Australia, and New Zealand. The first participant was screened on 17 July 2013. The last study visit occurred on 14 May 2015.
Pre-assignment Details: A total of 1255 participants were screened of which 599 participants were randomized into the study and only 594 participants were treated.
Period: Period 1 (Baseline up to Week 12)
Arm/Group | Placebo | GLPG0634 50 mg QD | GLPG0634 100 mg QD | GLPG0634 200 mg QD | GLPG0634 25 mg BID | GLPG0634 50 mg BID | GLPG0634 100 mg BID
Started | 86 | 82 | 85 | 86 | 86 | 85 | 84
Completed | 83 | 76 | 78 | 80 | 77 | 80 | 83
Not Completed | 3 | 6 | 7 | 6 | 9 | 5 | 1
Not completed — Withdrawal by Subject | 2 | 2 | 3 | 4 | 3 | 0 | 0
Not completed — Other | 1 | 0 | 1 | 1 | 3 | 3 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 2 | 3 | 1 | 2 | 1 | 0
Not completed — Adverse event and treatment failure | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Non-compliance with the study procedures | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 1 | 0
Period: Period 2 (Week 13 to Week 24)
Arm/Group | Placebo | GLPG0634 50 mg QD | GLPG0634 100 mg QD | GLPG0634 200 mg QD | GLPG0634 25 mg BID | GLPG0634 50 mg BID | GLPG0634 100 mg BID
Started | 53 (Nonresponders from Placebo group moved to 100 mg QD(15 participants) and 50 mg BID(15 participants).) | 57 (Nonresponders from 50 mg QD group moved to 100 mg QD group (19 participants).) | 112 (Nonresponders from Placebo(15 participants) and 50 mg QD (19 participants) moved to 100 mg QD group.) | 80 | 60 (Nonresponders from 25 mg BID group moved to 50 mg BID group (17 participants).) | 112 (Nonresponders from Placebo(15 participants) and 25 mg BID(17 participants) moved to 50 mg BID group.) | 83
Completed | 50 | 55 | 104 | 78 | 57 | 109 | 80
Not Completed | 3 | 2 | 8 | 2 | 3 | 3 | 3
Not completed — Withdrawal by Subject | 1 | 1 | 2 | 0 | 1 | 0 | 0
Not completed — Adverse event and treatment failure | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Non compliance with study medication | 0 | 0 | 2 | 0 | 0 | 1 | 0
Not completed — Treatment failure | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 3 | 2 | 1 | 1 | 3
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who were randomized and received at least one dose of study medication.
Groups:
- Placebo: Participants received GLPG0634 matching placebo capsules, orally, BID during Weeks 1 to 12. Participants who were responders (having at least 20 percent% improvement on TJC68 and SJC66) remained on placebo while nonresponders were re-randomized to GLPG0634 100 mg QD or 50 mg BID during Weeks 13 to 24.
- Total: Total of all reporting groups
Arm/Group | Placebo | GLPG0634 50 mg QD | GLPG0634 100 mg QD | GLPG0634 200 mg QD | GLPG0634 25 mg BID | GLPG0634 50 mg BID | GLPG0634 100 mg BID | Total
Number analyzed (Participants) | 86 | 82 | 85 | 86 | 86 | 85 | 84 | 594
Age, Continuous [Mean (Full Range); unit: years] | 52 [18 to 84] | 52.8 [20 to 77] | 52.3 [20 to 79] | 54.8 [19 to 75] | 52.4 [24 to 79] | 55.4 [21 to 78] | 53.9 [22 to 76] | 53.4 [18 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 69 | 65 | 74 | 68 | 65 | 70 | 481
  Male | 16 | 13 | 20 | 12 | 18 | 20 | 14 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37 | 37 | 33 | 33 | 37 | 30 | 38 | 245
  Not Hispanic or Latino | 49 | 45 | 52 | 53 | 49 | 55 | 46 | 349
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 3
  White | 59 | 61 | 62 | 67 | 63 | 65 | 66 | 443
  More than one race | 26 | 21 | 22 | 18 | 23 | 19 | 17 | 146
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rheumatoid Arthritis (RA) duration [Mean (Full Range); unit: years] | 8.21 [0.5 to 36.5] | 7.21 [0.6 to 21.3] | 7.67 [0.6 to 32.6] | 8.51 [0.5 to 34.5] | 8.88 [0.5 to 30.1] | 7.79 [0.5 to 28.8] | 9.74 [0.5 to 43.2] | 8.29 [0.5 to 43.2]
C-reactive protein (CRP) at Baseline [Mean (Full Range); unit: milligram per liter (mg/L)] | 16.25 [1 to 84.5] | 27.71 [1 to 158.7] | 24.54 [1 to 140.7] | 27.1 [1 to 140.9] | 26.01 [1.2 to 157.3] | 24.6 [1 to 113.4] | 26.86 [1 to 129.4] | 24.70 [1 to 158.7]
Corrected tender joint count based on 68 joints (TJC68) at Baseline [Mean (Full Range); unit: joint count] — 68 joints were assessed for tenderness and joints are classified as tender/not tender giving a total possible tender joint count score of 0 to 68.
  joint count | 24.984 [8 to 60] | 24.907 [8 to 64] | 25.319 [8 to 68] | 28.843 [8 to 68] | 25.427 [8 to 64] | 27.158 [8 to 66] | 25.946 [7 to 61] | 26.091 [7 to 68]
Corrected swollen joint count based on 66 joints (SJC66) at Baseline [Mean (Full Range); unit: joint count] — 66 joints were assessed for swelling and joints are classified as swollen/not swollen giving a total possible swollen joint count score of 0 to 66.
  joint count | 16.13 [6 to 48] | 17.023 [6 to 66] | 16.31 [6 to 54] | 17.355 [6 to 58] | 15.663 [6 to 40] | 17.534 [6 to 62] | 16.356 [6 to 48] | 16.622 [6 to 66]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving an American College of Rheumatology (ACR) 20 Response at Week 12
Description: The American College of Rheumatology (ACR) response is a measurement of improvement in multiple disease assessment criteria. The ACR20 response is defined as: 1) ≥ 20% improvement from baseline in SJC66, and 2) ≥ 20% improvement from baseline in tender TJC68, and 3) ≥ 20% improvement from baseline in at least 3 of the following 5 items: 1. Pain visual analog scale (VAS) (taken from the Health Assessment Questionnaire - Disability Index [HAQ-DI]), 2. Patient's Global Assessment of Disease Activity VAS, 3. Physician's Global Assessment of Disease Activity VAS, 4. Total HAQ-DI score, and 5. CRP. Non-responder imputation was used (ie, to impute a missing response, the participant was assumed to be a non-responder).
Time Frame: Week 12
Population: Intent-to-treat (ITT) population included all participants in the safety population who had post-randomization data for at least one efficacy parameter.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | GLPG0634 50 mg QD | GLPG0634 100 mg QD | GLPG0634 200 mg QD | GLPG0634 25 mg BID | GLPG0634 50 mg BID | GLPG0634 100 mg BID
Number analyzed (Participants) | 86 | 82 | 85 | 86 | 86 | 85 | 84
percentage of participants | 44.2 | 56.1 | 63.5 | 68.6 | 57 | 60 | 78.6
Statistical Analysis 1: Comparison: Placebo vs GLPG0634 50 mg QD; Pairwise comparisons of each group vs. the placebo group using a logistic regression model with factors treatment group, geographical region, and prior use of biologics; Test type: Superiority; p = 0.1236, Regression, Logistic; P-value has been corrected for multiplicity according to Hommel's closed-testing method; Difference in percentage rates = 11.9, 95% CI 2-sided [-3.1 to 26.9]
Statistical Analysis 2: Comparison: Placebo vs GLPG0634 100 mg QD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0435, Regression, Logistic — P-value has been corrected for multiplicity according to Hommel's closed-testing method; Difference in percentage rates = 19.3, 95% CI 2-sided [4.7 to 34]
Statistical Analysis 3: Comparison: Placebo vs GLPG0634 200 mg QD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0068, Regression, Logistic — P-value has been corrected for multiplicity according to Hommel's closed-testing method; Difference in percentage rates = 24.4, 95% CI 2-sided [10.1 to 38.8]
Statistical Analysis 4: Comparison: Placebo vs GLPG0634 25 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.1236, Regression, Logistic — P-value has been corrected for multiplicity according to Hommel's closed-testing method; Difference in percentage rates = 12.8, 95% CI 2-sided [-2 to 27.6]
Statistical Analysis 5: Comparison: Placebo vs GLPG0634 50 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.1056, Regression, Logistic — P-value has been corrected for multiplicity according to Hommel's closed-testing method; Difference in percentage rates = 15.8, 95% CI 2-sided [1 to 30.6]
Statistical Analysis 6: Comparison: Placebo vs GLPG0634 100 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Logistic — P-value has been corrected for multiplicity according to Hommel's closed-testing method; Difference in percentage rates = 34.4, 95% CI 2-sided [20.7 to 48.1]

2. Secondary Outcome: Percentage of Participants Achieving an ACR20 Response at Week 24
Description: ACR20 response was defined as: 1) ≥ 20% improvement from baseline in SJC66, and 2) ≥ 20% improvement from baseline in TJC68, and 3) ≥ 20% improvement from baseline in at least 3 of the following 5 items: 1. Pain VAS (taken from the HAQ-DI), 2. Patient's Global Assessment of Disease Activity VAS, 3. Physician's Global Assessment of Disease Activity VAS, 4. Total HAQ-DI score, and 5. CRP. Non-responder imputation was used.
Time Frame: Week 24
Population: ITT population. Participants who switched treatment at Week 12 were handled as if they discontinued at Week 12.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | GLPG0634 50 mg QD | GLPG0634 100 mg QD | GLPG0634 200 mg QD | GLPG0634 25 mg BID | GLPG0634 50 mg BID | GLPG0634 100 mg BID
Number analyzed (Participants) | 86 | 82 | 85 | 86 | 86 | 85 | 84
percentage of participants | 41.9 | 54.9 | 61.2 | 73.3 | 55.8 | 60 | 79.8

3. Secondary Outcome: Percentage of Participants Achieving an ACR50 Response at Weeks 1, 2, 4, 8, 12, and 24
Description: ACR50 response was defined as: 1) ≥ 50% improvement from baseline in SJC66, and 2) ≥ 50% improvement from baseline in TJC68, and 3) ≥ 50% improvement from baseline in at least 3 of the following 5 items: 1. Pain VAS (taken from the HAQ-DI) 2. Patient's Global Assessment of Disease Activity VAS 3. Physician's Global Assessment of Disease Activity VAS 4. Total HAQ-DI score 5. CRP. Non-responder imputation was used.
Time Frame: Weeks 1, 2, 4, 8, 12, and 24
Population: ITT population. Participants who switched treatment at Week 12 were handled as if they discontinued at Week 12.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | GLPG0634 50 mg QD | GLPG0634 100 mg QD | GLPG0634 200 mg QD | GLPG0634 25 mg BID | GLPG0634 50 mg BID | GLPG0634 100 mg BID
Number analyzed (Participants) | 86 | 82 | 85 | 86 | 86 | 85 | 84
percentage of participants
  Week 1 | 1.2 | 2.4 | 4.7 | 4.7 | 3.5 | 7.1 | 7.1
  Week 2 | 5.8 | 7.3 | 20 | 10.5 | 7 | 11.8 | 21.4
  Week 4 | 7 | 13.4 | 32.9 | 17.4 | 15.1 | 18.8 | 34.5
  Week 8 | 12.8 | 26.8 | 35.3 | 33.7 | 25.6 | 34.1 | 45.2
  Week 12 | 15.1 | 32.9 | 37.6 | 43 | 27.9 | 34.1 | 54.8
  Week 24 | 16.3 | 35.4 | 47.1 | 50 | 34.9 | 35.3 | 54.8

4. Secondary Outcome: Percentage of Participants Achieving an ACR70 Response at Weeks 1, 2, 4, 8, 12, and 24
Description: ACR70 response: 1) ≥ 70% improvement from baseline in SJC66, and 2) ≥ 70% improvement from baseline in TJC68, and 3) ≥ 70% improvement from baseline in at least 3 of the following 5 items: 1. Pain VAS (taken from the HAQ-DI), 2. Patient's Global Assessment of Disease Activity VAS, 3. Physician's Global Assessment of Disease Activity VAS, 4. Total HAQ-DI score, and 5. CRP. Non-responder imputation was used.
Time Frame: Weeks 1, 2, 4, 8, 12, and 24
Population: ITT population. Participants who switched treatment at Week 12 were handled as if they discontinued at Week 12.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | GLPG0634 50 mg QD | GLPG0634 100 mg QD | GLPG0634 200 mg QD | GLPG0634 25 mg BID | GLPG0634 50 mg BID | GLPG0634 100 mg BID
Number analyzed (Participants) | 86 | 82 | 85 | 86 | 86 | 85 | 84
percentage of participants
  Week 1 | 1.2 | 0 | 0 | 1.2 | 1.2 | 2.4 | 4.8
  Week 2 | 1.2 | 2.4 | 7.1 | 5.8 | 2.3 | 5.9 | 3.6
  Week 4 | 3.5 | 7.3 | 14.1 | 4.7 | 5.8 | 9.4 | 10.7
  Week 8 | 7 | 11 | 23.5 | 18.6 | 9.3 | 14.1 | 27.4
  Week 12 | 8.1 | 15.9 | 21.2 | 24.4 | 14 | 18.8 | 31
  Week 24 | 9.3 | 22 | 32.9 | 29.1 | 20.9 | 23.5 | 39.3

5. Secondary Outcome: ACR N% Improvement (ACR-N) Response at Weeks 1, 2, 4, 8, 12, and 24
Description: The ACR-N is the smallest percentage improvement in swollen and tender joints and the median of the remaining 5 core parameters, and is expected to be more sensitive to change than the ACR20, ACR50 or ACR70. It is a number varying between 0 and 100, with higher numbers indicating less severity of symptoms. Last observation carried forward (LOCF) algorithm was used (ie, to impute a missing value, the last preceding nonmissing value was used).
Time Frame: Weeks 1, 2, 4, 8, 12, and 24
Population: ITT population with available data were analyzed. Participants who switched treatment at Week 12 were handled as if they discontinued at Week 12.
Measure: Mean (Standard Error); unit: percentage of improvement
Arm/Group | Placebo | GLPG0634 50 mg QD | GLPG0634 100 mg QD | GLPG0634 200 mg QD | GLPG0634 25 mg BID | GLPG0634 50 mg BID | GLPG0634 100 mg BID
Number analyzed (Participants) | 84 | 82 | 80 | 86 | 83 | 85 | 82
percentage of improvement
  Week 1 | 9.27 (1.519) | 10.31 (1.578) | 14.69 (2.04) | 14.25 (1.822) | 9.01 (1.603) | 11.36 (1.939) | 17.63 (2.206)
  Week 2 | 13.85 (1.949) | 16.36 (2.125) | 25.2 (1.986) | 22.61 (2.517) | 15.2 (2.063) | 20.01 (2.47) | 27.77 (2.606)
  Week 4 | 16.93 (2.332) | 21.08 (2.598) | 31.32 (3.354) | 27.45 (2.573) | 23.17 (2.668) | 26.37 (2.961) | 35.69 (2.861)
  Week 8 | 21.6 (2.644) | 30.16 (3.015) | 38.24 (3.484) | 37.88 (3.097) | 31.2 (2.845) | 33.4 (3.15) | 45.36 (3.246)
  Week 12 | 23.09 (2.911) | 34.03 (3.335) | 39.87 (3.449) | 42.1 (3.277) | 34.12 (3.144) | 35.86 (3.29) | 51.17 (3.379)
  Week 24 | 22.06 (2.846) | 37.13 (3.582) | 50.86 (3.645) | 50.4 (3.291) | 38.56 (3.384) | 40.5 (3.299) | 58.69 (3.204)

6. Secondary Outcome: Percentage of Participants With Disease Activity Score 28 Joints Corrected for CRP (DAS28 (CRP)) European League Against Rheumatism (EULAR) Response at Weeks 1, 2, 4, 8, 12, and 24
Description: DAS28 (CRP) was categorized into EULAR response categories (none, moderate, good) as follows: None = Actual DAS28 (CRP) ≤ 3.2, > 3.2 to ≤ 5.1, or > 5.1 AND Improvement in DAS28 (CRP) from baseline ≤ 6.0 or > 0.6 to ≤ 1.2; Moderate = Actual DAS28 (CRP) ≤ 3.2 AND Improvement in DAS28 (CRP) from baseline > 0.6 to ≤ 1.2, Actual DAS28 (CRP) > 3.2 to ≤ 5.1 or > 5.1 AND Improvement in DAS28 (CRP) from baseline > 1.2, or Actual DAS28 (CRP) > 3.2 to ≤ 5.1 AND Improvement in DAS28 (CRP) from baseline > 0.6 to ≤ 1.2; Good = Actual DAS28 (CRP) ≤ 3.2 AND Improvement in DAS28 (CRP) from baseline > 1.2. LOCF algorithm was used.
Time Frame: Weeks 1, 2, 4, 8, 12, and 24
Population: ITT population. Participants who switched treatment at Week 12 were handled as if they discontinued at Week 12.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | GLPG0634 50 mg QD | GLPG0634 100 mg QD | GLPG0634 200 mg QD | GLPG0634 25 mg BID | GLPG0634 50 mg BID | GLPG0634 100 mg BID
Number analyzed (Participants) | 86 | 82 | 85 | 86 | 86 | 85 | 84
percentage of participants
  Week 1: None | 73 | 61 | 58 | 42 | 63 | 64 | 40
  Week 1: Moderate | 21 | 38 | 35 | 55 | 34 | 32 | 49
  Week 1: Good | 6 | 1 | 7 | 3 | 3 | 5 | 11
  Week 2: None | 58 | 49 | 39 | 31 | 51 | 44 | 20
  Week 2: Moderate | 33 | 45 | 42 | 53 | 43 | 46 | 62
  Week 2: Good | 9 | 6 | 19 | 15 | 6 | 11 | 18
  Week 4: None | 56 | 44 | 29 | 16 | 37 | 35 | 15
  Week 4: Moderate | 34 | 46 | 40 | 65 | 44 | 42 | 61
  Week 4: Good | 10 | 10 | 31 | 19 | 19 | 22 | 24
  Week 8: None | 44 | 34 | 20 | 15 | 24 | 24 | 8
  Week 8: Moderate | 43 | 45 | 52 | 49 | 51 | 49 | 46
  Week 8: Good | 13 | 21 | 28 | 36 | 24 | 27 | 45
  Week 12: None | 41 | 33 | 18 | 8 | 28 | 15 | 7
  Week 12: Moderate | 45 | 44 | 48 | 55 | 44 | 56 | 43
  Week 12: Good | 14 | 23 | 34 | 37 | 28 | 28 | 50
  Week 24: None | 48 | 33 | 12 | 10 | 23 | 14 | 5
  Week 24: Moderate | 34 | 35 | 38 | 38 | 37 | 49 | 31
  Week 24: Good | 19 | 32 | 51 | 51 | 40 | 36 | 64

7. Secondary Outcome: Percentage of Participants Achieving ACR/EULAR Remission at Weeks 2, 4, 8, 12, and 24
Description: A participant's disease activity status can be defined as being in remission when scores on the TJC28, SJC28, CRP (actual value in mg/dL) and Patient Global Assessment of Disease Activity (cm) are all ≤ 1. Non-responder imputation was used.
Time Frame: Weeks 2, 4, 8, 12, and 24
Population: ITT population. Participants who switched treatment at Week 12 were handled as if they discontinued at Week 12.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | GLPG0634 50 mg QD | GLPG0634 100 mg QD | GLPG0634 200 mg QD | GLPG0634 25 mg BID | GLPG0634 50 mg BID | GLPG0634 100 mg BID
Number analyzed (Participants) | 86 | 82 | 85 | 86 | 86 | 85 | 84
percentage of participants
  Week 2 | 0 | 0 | 3.5 | 0 | 0 | 0 | 1.2
  Week 4 | 1.2 | 1.2 | 1.2 | 2.3 | 0 | 0 | 2.4
  Week 8 | 1.2 | 3.7 | 3.5 | 3.5 | 1.2 | 1.2 | 3.6
  Week 12 | 3.5 | 3.7 | 3.5 | 5.8 | 4.7 | 4.7 | 9.5
  Week 24 | 1.2 | 11 | 8.2 | 11.6 | 5.8 | 3.5 | 19

8. Secondary Outcome: Change From Baseline in Simplified Disease Activity Index (SDAI) at Weeks 1, 2, 4, 8, 12, and 24
Description: The SDAI is the numerical sum of 5 outcome parameters: TJC28, SJC28, Patient Global Assessment of Disease Activity (in cm), Physician's Global Assessment of Disease Activity (in cm), and CRP (mg/dL). The SDAI was categorized as follows:
  • High disease activity: SDAI > 26 • Moderate disease activity: 11 to 26 • Low disease activity: 3.3 to 11 • Remission: ≤ 3.3. LOCF algorithm was used. The SDAI total score ranges from 0 to approximately 86.
Time Frame: Baseline and Weeks 1, 2, 4, 8, 12, and 24
Population: as for outcome 5
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | GLPG0634 50 mg QD | GLPG0634 100 mg QD | GLPG0634 200 mg QD | GLPG0634 25 mg BID | GLPG0634 50 mg BID | GLPG0634 100 mg BID
Number analyzed (Participants) | 86 | 82 | 85 | 86 | 86 | 85 | 84
units on a scale
  Baseline | 43.756 (1.2717) | 43.77 (1.3499) | 45.42 (1.3909) | 45.611 (1.3362) | 43.951 (1.3224) | 44.794 (1.4043) | 44.542 (1.3097)
  Change at Week 1: number analyzed (Participants) | 86 | 82 | 85 | 86 | 85 | 85 | 84
  Change at Week 1 | -8.3 (1.25) | -8 (1.14) | -12.2 (1.45) | -12.8 (1.29) | -8.2 (1.17) | -10 (1.22) | -14.5 (1.31)
  Change at Week 2: number analyzed (Participants) | 86 | 82 | 85 | 86 | 85 | 85 | 84
  Change at Week 2 | -11.4 (1.45) | -12.5 (1.46) | -18.6 (1.64) | -16.4 (1.35) | -13.4 (1.29) | -15.1 (1.43) | -20.3 (1.35)
  Change at Week 4: number analyzed (Participants) | 86 | 82 | 85 | 86 | 85 | 85 | 84
  Change at Week 4 | -13.1 (1.47) | -16.3 (1.64) | -22.7 (1.78) | -22.2 (1.28) | -17.8 (1.44) | -19.3 (1.74) | -24.9 (1.54)
  Change at Week 8: number analyzed (Participants) | 86 | 82 | 85 | 86 | 85 | 85 | 84
  Change at Week 8 | -16.3 (1.64) | -20.1 (1.86) | -24.6 (1.57) | -25.9 (1.57) | -22.2 (1.68) | -23.2 (1.8) | -29.2 (1.58)
  Change at Week 12: number analyzed (Participants) | 86 | 82 | 85 | 86 | 85 | 85 | 84
  Change at Week 12 | -16.3 (1.84) | -21 (1.84) | -25.2 (1.69) | -27.2 (1.55) | -22.3 (1.71) | -24.5 (1.87) | -30.6 (1.57)
  Change at Week 24: number analyzed (Participants) | 86 | 82 | 85 | 86 | 85 | 85 | 84
  Change at Week 24 | -15.8 (2) | -22.8 (2.07) | -30.1 (1.66) | -31 (1.66) | -24.9 (1.85) | -27.9 (2) | -34.4 (1.47)

9. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) at Weeks 1, 2, 4, 8, 12, and 24
Description: The CDAI is the SDAI modified to exclude CRP and is the sum of the 4 outcome parameters: TJC28, SJC28, Patient Global Assessment of Disease Activity (in cm), and Physician's Global Assessment of Disease Activity (in cm). The CDAI was be categorized as follows: • High disease activity: > 22 • Moderate disease activity: 10 to 22 • Mild disease activity: 2.8 to 10 • Remission: ≤ 2.8. LOCF algorithm was used. The CDAI total score ranges from 0 to approximately 76.
Time Frame: Baseline and Weeks 1, 2, 4, 8, 12, and 24
Population: as for outcome 5
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | GLPG0634 50 mg QD | GLPG0634 100 mg QD | GLPG0634 200 mg QD | GLPG0634 25 mg BID | GLPG0634 50 mg BID | GLPG0634 100 mg BID
Number analyzed (Participants) | 86 | 82 | 85 | 86 | 86 | 85 | 84
units on a scale
  Baseline | 42.131 (1.236) | 40.999 (1.2104) | 42.966 (1.3014) | 42.901 (1.2844) | 41.347 (1.2442) | 42.333 (1.3186) | 41.856 (1.2462)
  Change at Week 1: number analyzed (Participants) | 86 | 82 | 85 | 86 | 85 | 85 | 84
  Change at Week 1 | -8.5 (1.23) | -7.2 (1.09) | -11.1 (1.38) | -11.1 (1.22) | -7.3 (1.14) | -9 (1.15) | -12.8 (1.27)
  Change at Week 2: number analyzed (Participants) | 86 | 82 | 85 | 86 | 85 | 85 | 84
  Change at Week 2 | -11.6 (1.43) | -11.7 (1.39) | -17.3 (1.58) | -14.6 (1.29) | -12.4 (1.26) | -14 (1.38) | -18.4 (1.31)
  Change at Week 4: number analyzed (Participants) | 86 | 82 | 85 | 86 | 85 | 85 | 84
  Change at Week 4 | -13.3 (1.42) | -15.2 (1.54) | -21.4 (1.71) | -20.4 (1.24) | -17.1 (1.35) | -18 (1.71) | -22.8 (1.51)
  Change at Week 8: number analyzed (Participants) | 86 | 82 | 85 | 86 | 85 | 85 | 84
  Change at Week 8 | -16.4 (1.58) | -18.9 (1.78) | -23.4 (1.52) | -24.2 (1.15) | -21.1 (1.67) | -21.9 (1.75) | -27.1 (1.53)
  Change at Week 12: number analyzed (Participants) | 86 | 82 | 85 | 86 | 85 | 85 | 84
  Change at Week 12 | -16.6 (1.84) | -19.7 (1.77) | -23.8 (1.66) | -25.5 (1.5) | -21.3 (1.65) | -23.2 (1.81) | -28.5 (1.49)
  Change at Week 24: number analyzed (Participants) | 86 | 82 | 85 | 86 | 85 | 85 | 84
  Change at Week 24 | -16 (1.95) | -21.3 (1.97) | -28.6 (1.63) | -29.4 (1.5) | -23.8 (1.75) | -26.7 (1.9) | -32.4 (1.39)

10. Secondary Outcome: Change From Baseline in Quality of Life Using the Functional Assessment of Chronic Illness Therapy (FACIT) at Weeks 4, 12, and 24
Description: FACIT-Fatigue scale is a 13-item questionnaire, each scored on a 5-point scale: 0 (Not at all) to 4 (Very much). The larger the participant's response to the questions (with the exception of 2 negatively stated that are scored reversely), the greater the fatigue. The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score), with a higher score indicating a better quality of life. LOCF algorithm was used.
Time Frame: Baseline and Weeks 4, 12, and 24
Population: as for outcome 5
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | GLPG0634 50 mg QD | GLPG0634 100 mg QD | GLPG0634 200 mg QD | GLPG0634 25 mg BID | GLPG0634 50 mg BID | GLPG0634 100 mg BID
Number analyzed (Participants) | 86 | 82 | 85 | 86 | 86 | 85 | 84
units on a scale
  Baseline | 26.2 (1.09) | 26.2 (1.1) | 26.6 (1.06) | 25.2 (1.25) | 28.1 (1.18) | 26.2 (1.04) | 25.6 (1.25)
  Change at Week 4: number analyzed (Participants) | 86 | 82 | 84 | 86 | 86 | 85 | 83
  Change at Week 4 | 4.9 (1.06) | 4.4 (1.11) | 9.1 (1.14) | 8.5 (1.23) | 4.5 (1.06) | 6.6 (0.88) | 9.9 (0.97)
  Change at Week 12: number analyzed (Participants) | 86 | 82 | 84 | 86 | 86 | 85 | 83
  Change at Week 12 | 5.6 (1.06) | 7.6 (1.26) | 9.5 (1.21) | 11.4 (1.37) | 6.9 (1.12) | 8.4 (1.08) | 11.3 (1.25)
  Change at Week 24: number analyzed (Participants) | 86 | 82 | 84 | 86 | 86 | 85 | 83
  Change at Week 24 | 6 (1.04) | 7.9 (1.21) | 11.1 (1.2) | 11.6 (1.33) | 7.7 (1.17) | 9 (1.04) | 12.8 (1.36)

11. Secondary Outcome: Change From Baseline in Quality of Life Using the Short Form-36 (SF-36) Scores at Weeks 4, 12, and 24
Description: The SF-36 is a 36-item questionnaire measuring 8 domains (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health). Each domain score ranges from 0 (worst) to 100 (best), with higher scores reflecting better health-related functional status. Two summary scale scores were computed based on weighted combinations of the 8 domain scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). LOCF algorithm was used.
Time Frame: Baseline and Weeks 4, 12, and 24
Population: as for outcome 5
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | GLPG0634 50 mg QD | GLPG0634 100 mg QD | GLPG0634 200 mg QD | GLPG0634 25 mg BID | GLPG0634 50 mg BID | GLPG0634 100 mg BID
Number analyzed (Participants) | 86 | 82 | 85 | 86 | 86 | 85 | 84
units on a scale
  PCS at Baseline | 32.999 (0.7121) | 32.691 (0.7474) | 31.636 (0.7926) | 31.625 (0.6355) | 31.364 (0.6858) | 31.332 (0.726) | 32.249 (0.7844)
  PCS Change at Week 4: number analyzed (Participants) | 86 | 82 | 84 | 86 | 86 | 85 | 83
  PCS Change at Week 4 | 3 (0.65) | 4.1 (0.88) | 6.1 (0.98) | 6.4 (0.87) | 5 (0.69) | 4.2 (0.8) | 7.2 (0.77)
  PCS Change at Week 12: number analyzed (Participants) | 86 | 82 | 84 | 86 | 86 | 85 | 83
  PCS Change at Week 12 | 3.2 (0.74) | 6.7 (1) | 8.4 (0.93) | 8.9 (0.9) | 7.5 (0.92) | 7.1 (0.96) | 10.5 (0.98)
  PCS Change at Week 24: number analyzed (Participants) | 86 | 82 | 84 | 86 | 86 | 85 | 83
  PCS Change at Week 24 | 2.8 (0.75) | 7.3 (1.02) | 9.9 (1.09) | 9.7 (0.99) | 7.8 (0.85) | 7.9 (0.91) | 11.6 (1.1)
  MCS at Baseline | 42.849 (1.0861) | 42.199 (1.2581) | 43.953 (1.1118) | 41.362 (1.1427) | 45.527 (1.288) | 44.748 (1.228) | 42.059 (1.2898)
  MCS at Week 4: number analyzed (Participants) | 86 | 82 | 84 | 86 | 86 | 85 | 83
  MCS at Week 4 | 3 (0.92) | 3.4 (0.91) | 4.9 (0.85) | 5.4 (0.98) | 2.4 (0.78) | 2.7 (0.84) | 5.6 (0.92)
  MCS at Week 12: number analyzed (Participants) | 86 | 82 | 84 | 86 | 86 | 85 | 83
  MCS at Week 12 | 4.3 (1.05) | 4.4 (1.11) | 5.1 (0.96) | 8.1 (1.17) | 3.5 (0.97) | 3.1 (1.02) | 6.2 (0.98)
  MCS at Week 24: number analyzed (Participants) | 86 | 82 | 84 | 86 | 86 | 85 | 83
  MCS at Week 24 | 4.7 (0.96) | 4.3 (1.04) | 6.7 (0.91) | 7.2 (1.12) | 3.8 (0.96) | 3.5 (1.01) | 7.1 (1.21)

ADVERSE EVENTS:
Time Frame: Baseline through end of study drug treatment (average exposure: 160.7 days) plus 10 days
Description: Nonresponders from Placebo (15 participants), 50 mg QD (19 participants) moved to 100 mg QD group and nonresponders from Placebo (15 participants) and 25 mg BID (17 participants) moved to 50 mg BID group from Week 13 to Week 24.
Arm/Group | Placebo | GLPG0634 50 mg QD | GLPG0634 100 mg QD | GLPG0634 200 mg QD | GLPG0634 25 mg BID | GLPG0634 50 mg BID | GLPG0634 100 mg BID
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/82 | 0/119 | 0/86 | 0/86 | 0/117 | 1/84
Serious Adverse Events (participants affected / at risk) | 4/86 | 0/82 | 4/119 | 2/86 | 2/86 | 0/117 | 3/84
Other Adverse Events (participants affected / at risk) | 11/86 | 23/82 | 13/119 | 21/86 | 23/86 | 22/117 | 15/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=86) | GLPG0634 50 mg QD (N=82) | GLPG0634 100 mg QD (N=119) | GLPG0634 200 mg QD (N=86) | GLPG0634 25 mg BID (N=86) | GLPG0634 50 mg BID (N=117) | GLPG0634 100 mg BID (N=84)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abortion spontaneous complete (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Inflammation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Diabetic gangrene (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intervertebral discitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=86) | GLPG0634 50 mg QD (N=82) | GLPG0634 100 mg QD (N=119) | GLPG0634 200 mg QD (N=86) | GLPG0634 25 mg BID (N=86) | GLPG0634 50 mg BID (N=117) | GLPG0634 100 mg BID (N=84)
Hypertension (Vascular disorders) | 2 | 3 | 6 | 4 | 3 | 4 | 1
Headache (Nervous system disorders) | 4 | 1 | 1 | 6 | 6 | 3 | 2
Nausea (Gastrointestinal disorders) | 3 | 7 | 0 | 3 | 3 | 3 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 6 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 5 | 2 | 1 | 4
Gastroenteritis (Infections and infestations) | 0 | 1 | 1 | 2 | 5 | 2 | 1
Nasopharyngitis (Infections and infestations) | 4 | 8 | 3 | 3 | 4 | 2 | 4
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 2 | 4 | 4 | 6 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must review and approve any results of the study or abstracts for professional meetings prepared by the investigator(s). Published data must not compromise the objectives of the study. Data from individual study centers in multicenter studies must not be published separately.

DOCUMENTS (2):
  • Study Protocol (2014-05-27): https://cdn.clinicaltrials.gov/large-docs/74/NCT01888874/Prot_000.pdf
  • Statistical Analysis Plan (2015-06-18): https://cdn.clinicaltrials.gov/large-docs/74/NCT01888874/SAP_001.pdf